CLINICAL TRIAL: NCT04809415
Title: Influence of Power and Wavelength on Photobiomodulation Therapy for Muscle Performance in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rinaldo Roberto de Jesus Guirro, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: DifPower
Record Dates: First submitted 2021-03-17; First posted 2021-03-22 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Low Level Laser Therapy; Photobiomodulation; Performance; Sport
Keywords: Physical Therapy; Photobiomodulation; Muscle Strength; Power; Athletic Performance
MeSH Terms: interventions — Low-Level Light Therapy; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sham Group (G-S) (Sham Comparator): The LED blanket will be positioned across the quadriceps and hamstring bilaterally, however, there will be no light emission. However, the volunteer will perform the strength training protocol.
  Interventions: Other: Sham
- 300J Infrared Blanket LED Group (Blanket-300J) (Experimental): The LED blanket with a wavelength of 940nm, energy of 300J, will be applied across the quadriceps and hamstrings bilaterally, just before the strength training protocol.
  Interventions: Other: Photobiomodulation
- 300J Infrared Cluster LED Group (Cluster-300J) (Experimental): The LED Cluster with a wavelength of 850 nm, energy of 300 J, will be applied to the quadriceps (5 points) and hamstrings (5 points), bilaterally, just before the strength training protocol.
  Interventions: Other: Photobiomodulation

INTERVENTIONS:
Other: Photobiomodulation — Photobiomodulation consists of irradiation by light in order to achieve photochemical and photophysical outcomes.
  Arms: 300J Infrared Blanket LED Group (Blanket-300J); 300J Infrared Cluster LED Group (Cluster-300J)
Other: Sham — Simulation of the application of photobiomodulation therapy.
  Arms: Sham Group (G-S)

SUMMARY:
In recent years, photobiomodulation has been studied as a means of increasing muscle performance in athletes and healthy individuals. This is possible due to the physiological changes that photobiomodulation therapy can promote. Moreover, given a large number of existing studies on the subject, some directions for future research have been established. For example, future research was established, the relationship between power and time because with high power, it will achieve the same energy with shorter application times. However, irradiation may not be offered for the minimum recommended time. Therefore, this study aims to compare different powers and, consequently, different application times for muscle performance in healthy individuals. For this, 42 participants will be recruited, males between 18 to 40 years old, without recent musculoskeletal injury or cardiorespiratory problems. The participants will participate in 3 evaluations containing functional and physiological variables and ten training sessions of lower limbs with previous photobiomodulation therapy application, comparing devices with a power of 0.864W and 1.864W. 0.864W and 1.2W. Lower limbs training will be composed of stiff and squat exercises twice a week, for five weeks. In the pre- and post-intervention evaluations, the following parameters will be evaluated isokinetic apparatus, body composition, and functionality of the vertical jump. For data analysis, we will use a normality test to verify the distribution and statistical tests will be used for intra and intra and intergroup comparisons, considering two factors in the comparisons time and group. A significance level of 5% will be adopted.

DETAILED DESCRIPTION:
It is a blinded randomized clinical trial. The volunteers will undergo pre-evaluation, 5 weeks of training associated with the LED application, being distributed in two applications per week, and a re-evaluation 24 hours after the last application, totaling a total of approximately 7 weeks. Thus, on the first day (Pre-test) volunteers will be submitted to anthropometric evaluation and evaluation by bioimpedance for analysis of detailed body composition. Then, the maximum voluntary contraction test (CVM) will be performed on the isokinetic dynamometer, together with the electromyographic evaluation. Before and after the evaluation with the isokinetic dynamometer, thermography will be collected. Still, will be evaluated the vertical jump test after 15 minutes of passive rest.

After the initial evaluations, the researcher will go apply the respective interventions, which consist of applying LEDs all over the quadriceps and hamstring bilaterally, while the sham group (GS) will receive the LED application off, without the emission of light. The application will occur for five weeks and will occur twice weekly, on days spaced for at least 48 hours. The same will be done in conjunction with the lower limb strength training protocol. It is noteworthy that although the therapy follows the same energy values, two different pieces of equipment will be used, thus changing the wavelength, total power and power density, and the consequent coverage time and area.

The tests performed at the time of pre-application of the LED (Pre-test) will be reapplied in the same order 24 hours after the last application of the interventions. After seven days of the last application, the isokinetic evaluation, electromyography, and vertical jump evaluation will be performed. In addition, at the end of the second and fourth weeks, the volunteer will carry out an evaluation with the isokinetic dynamometer, electromyography, plethysmography, and thermography.

ELIGIBILITY:
Inclusion Criteria:

- healthy individuals;

Exclusion Criteria:

* musculoskeletal injury in the last three months;
* cardiovascular diseases;
* use of anabolic, anti-inflammatory and analgesic drugs 72 hours before the evaluations;
* use of alcohol and illicit drugs during the collection period;

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Difference of maximal voluntary contraction | 1 year
  The study was designed to detect a difference of maximal voluntary contraction between the groups, following the interventions

CONTACTS AND LOCATIONS:
Overall Officials: Carlos E Girasol, Student, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
The datas will be sharing in form of manuscript.

REFERENCES:
- [Background] American College of Sports Medicine. American College of Sports Medicine position stand. Progression models in resistance training for healthy adults. Med Sci Sports Exerc. 2009 Mar;41(3):687-708. doi: 10.1249/MSS.0b013e3181915670. PMID 19204579
- [Background] Ferraresi C, Beltrame T, Fabrizzi F, do Nascimento ES, Karsten M, Francisco Cde O, Borghi-Silva A, Catai AM, Cardoso DR, Ferreira AG, Hamblin MR, Bagnato VS, Parizotto NA. Muscular pre-conditioning using light-emitting diode therapy (LEDT) for high-intensity exercise: a randomized double-blind placebo-controlled trial with a single elite runner. Physiother Theory Pract. 2015 Jul;31(5):354-61. doi: 10.3109/09593985.2014.1003118. Epub 2015 Jan 14. PMID 25585514
- [Background] Anders JJ, Lanzafame RJ, Arany PR. Low-level light/laser therapy versus photobiomodulation therapy. Photomed Laser Surg. 2015 Apr;33(4):183-4. doi: 10.1089/pho.2015.9848. No abstract available. PMID 25844681